CLINICAL TRIAL: NCT04032340
Title: Companion Dog Impact on Loneliness and Social Link in Elderly Persons (≥ 75 Years Old) Living at Home : a Comparative Transversal Study
Brief Title: Companion Dog & Loneliness in Elderly Persons
Acronym: C-KDOG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation MUTAC (Unknown)
Responsible Party: Sponsor
Other Study IDs: AP-HP190493
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Elderly; Companion Dog; Home Based; Loneliness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly with a companion dog: elderly living at home with a dog consulting his family doctor
  Interventions: Other: dog presence
- Elderly without a companion dog: elderly living at home without a dog consulting his family doctor

INTERVENTIONS:
Other: dog presence — This project seeks to assess positive impacts of companion dog presence in elderly living at home ; to assess loneliness and isolement between eldlery with a companion dog and without, at home
  Groups: Elderly with a companion dog

SUMMARY:
Elderly may have problems to create personal connections or to have physical activities in their day- to - day life; loneliness and social isolation may increase fragility in this population. Companion dog presence favours social relations, affective feelings and physical exercises. On the other hand dog presence raises risk of falling and has a cost for its owner. This project seeks to assess positive impacts of companion dog presence in elderly living at home. This transdisciplinar study (general practionners, veterinarians, dog instructors, nurses, researchers) evaluates loneliness and social isolation between elderly with or without a companion dog at home.

Objective:To Evaluate the link between companion dog presence and loneliness in elderly persons living at home Method: An Observational, multicentric, transversal, national, comparative study (elderly with companion dog vs elderly without a dog). 200 subjects needed

ELIGIBILITY:
Inclusion Criteria:

* person aged ≥ 75years old
* living at home

Exclusion Criteria:

* bedridden person
* person accompanied by any animal, other than a dog
* EPHAD based (establishments providing care for the dependent elderly)
* comprehension or reading difficulties in french affecting study participation and scales assessment
* cognitive, mental ou psychic disorders
* person under legal protection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly (≥75 years old) living at home, with or without a companion dog, visiting their doctor
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
assessment of loneliness using Jong Gierveld scale (11items). | 5 to 10 days after inclusion visit
  emotional dimension (6items) social dimension (5items)

SECONDARY OUTCOMES:
social isolation | 5 to 10 days after inclusion visit
  Social Network Index french version (http://dx.doi.org/10.13072/midss.464)

CONTACTS AND LOCATIONS:
Overall Officials: FLORENCE CANOUI-POITRINE, MD-PHD, Principal Investigator — APHP CHU HENRI MONDOR

IPD SHARING:
Plan to Share IPD: No